CLINICAL TRIAL: NCT02202083
Title: The Comparison of Oxytocin Induced Labor and Cook Balloon Induced Labor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, qiang wei, Dr, West China Second University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: WCSH2014
Record Dates: First submitted 2014-06-22; First posted 2014-07-28 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Labor; Forced or Induced, Affecting Fetus or Newborn
Keywords: Oxytocin; Cook Balloon

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- oxytocin (Experimental): There are two groups. Acoording to the bishop score, one group uses the oxytocin , and the other uses the cook balloon.
  This group is term gestaion,with bishop score less than 6.
  Interventions: Other: Cook Balloon

INTERVENTIONS:
Other: Cook Balloon — There are two groups. Acoording to the bishop score, one group uses the oxytocin , and the other uses the cook balloon.
  This group is term gestaion,with bishop score less than 6.

SUMMARY:
Currently, the study about intervention on the induced abortion at trimester is so little. So, the investigators want to compare the safety and effectiveness of different induced labor.

DETAILED DESCRIPTION:
In this study , the investigators want to compare the safety and effectiveness of different induced labor. The safety and effectiveness such as the success rate of induced labor and the gestation outcome,etc.

ELIGIBILITY:
Inclusion Criteria:

* Gestation age ≥37week
* Single fetus
* No serious complications

Exclusion Criteria:

* Gestation age <37week
* Multiple fetus
* With serious complications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
The success rate of induced labor | one year

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, Dr, Study Director — West China second Hospital
Locations (1):
- West China Second Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- See also: this link is the official website of our hospital. — http://www.motherchildren.com